CLINICAL TRIAL: NCT06637787
Title: Prospective, Explorative, Research Study with Women to Investigate Menstruation Leakage At Night
Status: Active, not recruiting | Type: Observational
Sponsor: Essity Hygiene and Health AB (Industry)
Responsible Party: Sponsor
Other Study IDs: NOKTO
Record Dates: First submitted 2024-10-09; First posted 2024-10-15 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2024-10

CONDITIONS: Menstruation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Pads — A specially desigend pad is used to collect information about leakage and body movement at night.

SUMMARY:
The aim of this study is to investigate why and when menstruation leakages occur during sleep while using protective pads at night. Participants will be asked to use a specially designed pad during menstruation and to answer questions.

ELIGIBILITY:
Inclusion Criteria:

1. Women ≥ 18 years
2. Participant is mentally and physically able to participate in this study
3. Written informed consent to participate in this study
4. Participant with currently heavy menstruations regularly experiencing nocturnal leakages
5. Participant is a regular user of nocturnal menstruation pads
6. Participant is willing to use the prototype pad according to the protocol
7. Willingness to take picture of used pads and transfer to study sponsor anonymously during study duration
8. Available internet connection and device for taking pictures and data transfer (photo upload)
9. Underwear size M or L

Exclusion Criteria:

1. Known allergies or intolerances to one or several components of the study prototype
2. Participants without regular menstruation, pregnant or perimenopausal subjects
3. Participants not experiencing nocturnal leakages
4. Participants with pacemakers and/or implant defibrillator or having persons in the household that have a pacemaker and/or implant defibrillator

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with heavy menstruation
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-10-16 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Summary of leakage data of the menstruation pad in correlation with participats movements and position at leakage occasion. | 2025
  Leakage data and body movement will be assessed

SECONDARY OUTCOMES:
Evaluation of questionnaire to understand the sleeping pattern during period | 2025
  The answers received will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Essity Study site, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No